CLINICAL TRIAL: NCT03035656
Title: Effects of Intra-Operative Ropivaciane Epidural Injection on Post-Operative Outcomes Following Elective Lumbar Fusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Horizon Health Network (Other)
Responsible Party: Principal Investigator, Dr. neil Manson, Principal Investigator, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2016-2380
Record Dates: First submitted 2017-01-19; First posted 2017-01-30 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Pain, Postoperative
Keywords: Pain; analgesic; spinal fusion
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients are randomized into either the experimental arm (administration of Ropivaciane) or the control arm (administration of saline).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization of arms are conducted by the pharmacy department, and drug or saline preparation are prepared by the pharmacy department.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Administration of epidural Ropivaciane
  Interventions: Drug: Ropivacaine
- Control (Placebo Comparator): Administration of saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ropivacaine — Administration of Ropivaciane via epidural injection intra-operatively
  Arms: Experimental
Other: Saline — Administration of saline via epidural injection intra-operatively
  Arms: Control

SUMMARY:
The following is a double blinded, randomized controlled clinical trial to test the hypothesis that a single epidural injection of Ropivaciane® intra operatively will:1) Single intra-operative epidural injection of Ropivaciane® will result in decreased postoperative pain and opioid use in both minimally invasive (MIS) and open lumbar fusion patients; 2) Decreased postoperative pain will lead to improved clinical outcomes; and 3) Elucidate if there are differences in pain management between MIS and open surgical procedures. The proposed study will add novel information to current knowledge by 1) exploring of the effects of intra-operative single epidural injection analgesic on patients receiving MIS compared to open surgery, and 2) investigate potential immediate and short-term functional improvements gained from intra-operative single injection of Ropivaciane®.

DETAILED DESCRIPTION:
This double blinded, randomized clinical trial will test hypotheses by administering a single epidural injection prior to wound closure of either Ropivaciane® or saline.All pre-surgical activities and anesthesia will proceed as usual, with the addition of a single epidural injection immediately prior to wound closure 2 levels, or 10cm above the operated spinal level. Experimental groups will receive 0.2% Ropivaciane® (10 ml; dose shown to be effective without transient weakness), 9 and the control group will receive 0.9% saline solution (10 ml). Accurate placement into the space will be verified by the injection of contrast medium (iohexol, 180 mgl/ml) under fluoroscopic guidance. Epidural solutions will be prepared prior to surgery by pharmacy and coded; surgeons will administer according to the patient's code maintaining the double-blind procedure. It is important to note that treatment as usual differs between open and MIS cohorts. The question of interest is whether the addition of the epidural analgesic to current practices for each surgery type results in increased positive outcomes, whether this is due to synergistic effects or not. Following operative treatment, Foley Urinary catheter will be removed 24 hours post-operatively, unless otherwise clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Consenting participants undergoing elective 1-2 level lumbar fusion through the Canada East Spine Centre

Exclusion Criteria:

* History of severe respiratory, renal or hepatic disease
* Previous spine surgery
* Known allergy to local anaesthesia
* Those who experience dural tear during operative procedure

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | Administered 6 weeks pre-operatively, 2, 4, 8, 12, 24 and 48 hours post-operatively, 6 months post operatively, and 12 months post operatively
  Back and leg pain measured using the validated Numeric Rating Scales (NRS) for back and leg pain.

SECONDARY OUTCOMES:
Change in Disability | Administered 6 weeks pre-operatively, 6 and 12 months post-operatively
  Measurement of disability attributed to "back problem" using the validated Oswestry Disability Index (ODI).
Change in General Health | Administered 6 weeks pre-operatively, 6 and 12 months post-operatively
  Measurement of overall general health as measured by the validated Short Form General Health Survey (SF-12)
Change in Medication Use | Investigated 2, 4, 8, 12, 24 and 48 hours post-operatively.
  Medication used to control pain post-operatively as given by a qualified health professional while the patient is in hospital.

OTHER OUTCOMES:
Change in Ambulation | Investigated 2, 4, 8, 12, 24 and 48 hours post-operatively.
  The patient's ability to walk following surgery as measured using Ortho-Care Step Watch Activity Monitors (SAM) which will be attached to the patient's ankle during their stay in hospital.
Adverse Events | The total number of adverse events will be measured at the time of patient discharge, between 48 hours and 120 hours following surgical intervention
  Adverse Events (AEs) will be measured using the validated Spine Adverse

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Manson, MD FRCSC, Principal Investigator — Canada East Spine Centre; Horizon Health Network Department of Orthopaedic Surgery; Dalhousie University Faculty of Medicine Department of Surgery; Edward P Abraham, MD FRCSC, Principal Investigator — Canada East Spine Centre; Horizon Health Network Department of Orthopaedic Surgery; Dalhousie University Faculty of Medicine Department of Surgery

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Study results will be made available following data analysis.

REFERENCES:
- [Background] Raw DA, Beattie JK, Hunter JM. Anaesthesia for spinal surgery in adults. Br J Anaesth. 2003 Dec;91(6):886-904. doi: 10.1093/bja/aeg253. PMID 14633762
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Gessler F, Mutlak H, Tizi K, Senft C, Setzer M, Seifert V, Weise L. Postoperative patient-controlled epidural analgesia in patients with spondylodiscitis and posterior spinal fusion surgery. J Neurosurg Spine. 2016 Jun;24(6):965-70. doi: 10.3171/2015.8.SPINE15415. Epub 2016 Feb 5. PMID 26849711
- [Background] Hallivis R, Derksen TA, Meyr AJ. Peri-operative pain management. Clin Podiatr Med Surg. 2008 Jul;25(3):443-63; vii. doi: 10.1016/j.cpm.2008.02.006. PMID 18486854
- [Background] Sandkuhler J. Fear the pain. Lancet. 2002 Aug 10;360(9331):426. doi: 10.1016/S0140-6736(02)09683-6. No abstract available. PMID 12241712
- [Background] Carr DB, Goudas LC. Acute pain. Lancet. 1999 Jun 12;353(9169):2051-8. doi: 10.1016/S0140-6736(99)03313-9. PMID 10376632
- [Background] Breivik H. Postoperative pain management: why is it difficult to show that it improves outcome? Eur J Anaesthesiol. 1998 Nov;15(6):748-51. doi: 10.1097/00003643-199811000-00022. PMID 9884866
- [Background] Gottschalk A, Freitag M, Tank S, Burmeister MA, Kreil S, Kothe R, Hansen-Algenstedt N, Weisner L, Staude HJ, Standl T. Quality of postoperative pain using an intraoperatively placed epidural catheter after major lumbar spinal surgery. Anesthesiology. 2004 Jul;101(1):175-80. doi: 10.1097/00000542-200407000-00027. PMID 15220788
- [Background] Kang H, Jung HJ, Lee JS, Yang JJ, Shin HY, Song KS. Early postoperative analgesic effects of a single epidural injection of ropivacaine administered preoperatively in posterior lumbar interbody spinal arthrodesis: a pilot randomized controlled trial. J Bone Joint Surg Am. 2013 Mar 6;95(5):393-9. doi: 10.2106/JBJS.K.01729. PMID 23467861
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Chaney MA. Side effects of intrathecal and epidural opioids. Can J Anaesth. 1995 Oct;42(10):891-903. doi: 10.1007/BF03011037. PMID 8706199
- [Background] Kluba T, Hofmann F, Bredanger S, Blumenstock G, Niemeyer T. Efficacy of post-operative analgesia after posterior lumbar instrumented fusion for degenerative disc disease: a prospective randomized comparison of epidural catheter and intravenous administration of analgesics. Orthop Rev (Pavia). 2010 Mar 20;2(1):e9. doi: 10.4081/or.2010.e9. PMID 21808704
- [Background] Liu SS, Carpenter RL, Mackey DC, Thirlby RC, Rupp SM, Shine TS, Feinglass NG, Metzger PP, Fulmer JT, Smith SL. Effects of perioperative analgesic technique on rate of recovery after colon surgery. Anesthesiology. 1995 Oct;83(4):757-65. doi: 10.1097/00000542-199510000-00015. PMID 7574055
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Kehlet H, Dahl JB. The value of "multimodal" or "balanced analgesia" in postoperative pain treatment. Anesth Analg. 1993 Nov;77(5):1048-56. doi: 10.1213/00000539-199311000-00030. No abstract available. PMID 8105724
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591
- [Background] Mathiesen O, Dahl B, Thomsen BA, Kitter B, Sonne N, Dahl JB, Kehlet H. A comprehensive multimodal pain treatment reduces opioid consumption after multilevel spine surgery. Eur Spine J. 2013 Sep;22(9):2089-96. doi: 10.1007/s00586-013-2826-1. Epub 2013 May 17. PMID 23681498
- [Background] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Background] Woolf CJ. Recent advances in the pathophysiology of acute pain. Br J Anaesth. 1989 Aug;63(2):139-46. doi: 10.1093/bja/63.2.139. No abstract available. PMID 2669905
- [Background] Dworkin RH, O'Connor AB, Audette J, Baron R, Gourlay GK, Haanpaa ML, Kent JL, Krane EJ, Lebel AA, Levy RM, Mackey SC, Mayer J, Miaskowski C, Raja SN, Rice AS, Schmader KE, Stacey B, Stanos S, Treede RD, Turk DC, Walco GA, Wells CD. Recommendations for the pharmacological management of neuropathic pain: an overview and literature update. Mayo Clin Proc. 2010 Mar;85(3 Suppl):S3-14. doi: 10.4065/mcp.2009.0649. PMID 20194146
- [Background] Attal N, Cruccu G, Baron R, Haanpaa M, Hansson P, Jensen TS, Nurmikko T. EFNS guidelines on the pharmacological treatment of neuropathic pain: 2010 revision. Eur J Neurol. 2010 Sep;17(9):1113-e88. doi: 10.1111/j.1468-1331.2010.02999.x. Epub 2010 Apr 9. PMID 20402746
- [Background] Prasartritha T, Kunakornsawat S, Tungsiripat R, Jampa J, Throngnumchai R. A prospective randomized trial comparing epidural morphine through intraoperatively placed epidural catheter and intravenous morphine in major lumbar spinal surgery. J Spinal Disord Tech. 2010 Dec;23(8):e43-6. doi: 10.1097/BSD.0b013e3181cd3048. PMID 20924294
- [Background] Peters CL, Shirley B, Erickson J. The effect of a new multimodal perioperative anesthetic regimen on postoperative pain, side effects, rehabilitation, and length of hospital stay after total joint arthroplasty. J Arthroplasty. 2006 Sep;21(6 Suppl 2):132-8. doi: 10.1016/j.arth.2006.04.017. PMID 16950075
- [Background] Manchikanti L, Buenaventura RM, Manchikanti KN, Ruan X, Gupta S, Smith HS, Christo PJ, Ward SP. Effectiveness of therapeutic lumbar transforaminal epidural steroid injections in managing lumbar spinal pain. Pain Physician. 2012 May-Jun;15(3):E199-245. PMID 22622912
- [Background] Benyamin RM, Manchikanti L, Parr AT, Diwan S, Singh V, Falco FJ, Datta S, Abdi S, Hirsch JA. The effectiveness of lumbar interlaminar epidural injections in managing chronic low back and lower extremity pain. Pain Physician. 2012 Jul-Aug;15(4):E363-404. PMID 22828691
- [Background] Muller M, Burger C, Andermahr J, Mader K, Rangger C. [Spondylodiscitis after perioperative peridural catheter]. Anaesthesist. 2004 Dec;53(12):1189-94. doi: 10.1007/s00101-004-0764-3. German. PMID 15597159
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Vianin M. Psychometric properties and clinical usefulness of the Oswestry Disability Index. J Chiropr Med. 2008 Dec;7(4):161-3. doi: 10.1016/j.jcm.2008.07.001. PMID 19646379
- [Background] Luo X, George ML, Kakouras I, Edwards CL, Pietrobon R, Richardson W, Hey L. Reliability, validity, and responsiveness of the short form 12-item survey (SF-12) in patients with back pain. Spine (Phila Pa 1976). 2003 Aug 1;28(15):1739-45. doi: 10.1097/01.BRS.0000083169.58671.96. PMID 12897502